CLINICAL TRIAL: NCT05339035
Title: The Effect of Information, Motivation, Behavioral Skills Model-Based Motivational İnterview and Hippotherapy Program on Adolescents' Digital Game Addiction Levels
Brief Title: Digital Game Addiction in Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aslı Memis (Other)
Responsible Party: Sponsor-Investigator, Aslı Memis, lecturer, Amasya University
Organization: Amasya University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: lecturer
Record Dates: First submitted 2022-03-10; First posted 2022-04-21 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2022-04

CONDITIONS: Digital Technology; Behavior, Addictive; Adolescent; Motivation
Keywords: Digital Technology; Behavior, Addictive; Adolescent; Motivation
MeSH Terms: conditions — Behavior, Addictive

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- experimental group (Experimental): In the first stage, the participants will be trained according to the IMB model. In the second stage, 6 sessions of individual motivational interviews will be held for a total of 7 weeks. Finally, participants will be given hippotherapy 1 hour a week for 8 weeks.
  Interventions: Behavioral: Training based on IMB model, motivational interview technique, hippotherapy program
- control group (No Intervention): attempt will not be implemented.

INTERVENTIONS:
Behavioral: Training based on IMB model, motivational interview technique, hippotherapy program — In the first stage of the research, the "Digital Game Addiction Scale for Children" will be applied to the entire universe and participants with a digital game addiction score of 73 and above will be determined. According to the criteria of inclusion in the research, students will be informed and those who volunteer to participate in the study will be determined and listed. After the experimental and control groups are determined, the participants will be contacted and data collection forms will be applied. The students in the experimental group will be trained according to the IMB model, the students in the experimental group will be given a 6-session motivational interview program and the students will be taken to the hippotherapy program, which lasts 1 hour once a week for 8 weeks. Hippotherapy applications will be carried out at the horse farm in Amasya, accompanied by expert horsemen.
  Arms: experimental group

SUMMARY:
The research will be carried out on students studying at public secondary schools in the city center of Amasya. First of all, the digital game addiction levels of secondary school students who are randomly divided into experimental and control groups will be determined, and then students with digital game addiction will be included in the individual motivational interview program, which will last 6 sessions. In the last stage of the research, hippotherapy will be applied to the students 1 day a week for 8 weeks. The effect of motivational interviewing and hippoterain on digital game addiction will be investigated by pre-testing at the beginning of the research and post-testing at the end.

DETAILED DESCRIPTION:
The research was designed as a "pretest-posttest control group design type" quasi-experimental.

The population of the research consists of 6908 students enrolled in 35 secondary schools in Amasya city center and continuing their formal education. Among the students, 1730 students were determined as 5th Grade, 1763 as 6th Grade, 1754 as 7th Grade and 1661 as 8th Grade. Considering the intensity of the program, the 8th grade students who are preparing for the high school entrance exam are planned to be excluded from the study in order not to affect the study results negatively and considering that they will graduate from their schools during the follow-up process to be made at the end of the research. Private schools, secondary school students for the hearing impaired, 12 secondary school students in villages and towns will be excluded from the study, on the grounds that socioeconomic factors do not mislead the research results. There are a total of 4443 students studying in the 5th, 6th and 7th grades in 19 schools to be included in the study.

Power analysis (G*Power 3.1.9.7) was performed on the basis of a similar study performed before in calculating the sample size of the study. As a result of the power analysis, when the effect size was taken as 0.50 for the effect size, the sample number determined for 0.80 power and 0.05 margin of error was calculated as a total of 54 individuals, with a minimum of 27 individuals for each group. Considering that there may be sample losses during the research process, when 20% of the sample is added to each group, it is aimed to reach a total of 64 students, 32 students in the experimental group and 32 students in the control group.

2 secondary schools will be determined from a neighborhood in the city center of Amasya, and the experimental control separation of the schools will be determined by drawing lots. Schools will be selected from the same neighborhood so that there is no difference in socioeconomic levels between schools. In order to prevent the experimental and control groups from being influenced by each other, 2 different schools will be selected. The determined sample group will be randomly selected among the students with a digital game addiction score of 73 and above by using the "Digital Game Addiction Scale", and the research will be carried out with students who volunteer. Randomization will be done using the https://www.randomizer.org/ website.

Students in the experimental group will be trained according to the IMB model, motivational interviews will be made only with the experimental group, and the students will be included in the hippotherapy program, which lasts 1 hour once a week for 8 weeks. Hippotherapy applications will be carried out at the horse farm in Amasya, accompanied by expert horsemen.

ELIGIBILITY:
Inclusion Criteria:

* Being an official secondary school student
* Not having a physical disability
* Not doing sports/exercise for at least 30 minutes each time, 3 days a week
* Having a score of 73 or higher on the Digital Game Addiction Scale for Children
* Not riding a horse regularly
* Not afraid of horses and willing to ride

Exclusion Criteria:

* Being a private secondary school student
* Having a physical disability
* Do sports/exercise for at least 30 minutes each time, 3 days a week
* Having a score of 72 or less on the Digital Game Addiction Scale for Children
* Regular horseback riding
* Fear of horses and not willingness to ride

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 62 (Actual)
Dates: Start 2023-02-03 (Actual); Primary Completion 2023-12-26 (Actual); Study Completion 2024-04-22 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the 24-item Digital Game Addiction Scale score for Children at 8 weeks. | Baseline and Week 8
  The Digital Game Addiction Scale for Children is a validated, self-report tool that assesses the level of digital game addiction. The lowest score that can be obtained from the scale is "24" and the highest score is "120". In the grading of the scale scoring; It is evaluated as "1-24: Normal group, 25-48: Low risk group, 49-72 Risk group, 73-96 Dependent group, 97-120 Highly dependent group". Change = ( Week 8 score - Baseline score).

SECONDARY OUTCOMES:
Change from baseline in the 12-item Digital Game Addiction Awareness Scale score in 8 weeks. | Baseline and Week 8
  The Digital Game Addiction Awareness Scale is a validated, self-report tool that assesses the level of awareness of digital game addiction. The lowest score that can be obtained from the scale is "12" and the highest score is "60". Change = ( Week 8 score - Baseline score).

OTHER OUTCOMES:
Change in motivation to play digital games in the 19-item Digital Gaming Motivation Scale score at 8 weeks from baseline. | Baseline and Week 8
  The Digital Gaming Motivation Scale is a validated self-report tool that assesses the level of motivation to play digital games. The lowest score that can be obtained from the scale is "19" and the highest score is "95". Change = ( Week 8 score - Baseline score).
Change from baseline in the 41-item Social Support Assessment Scale score for Children and Adolescents at 8 weeks. | Baseline and Week 8
  The Social Support Rating Scale for Children and Adolescents is an approved self-report tool that assesses perceived social support level. The lowest score that can be obtained from the scale is "41" and the highest score is "205". Change = ( Week 8 score - Baseline score).
Change from baseline in the 18-item Digital Game Playing Attitude Scale score in 8 weeks. | Baseline and Week 8
  The Digital Gaming Attitude Scale is a validated, self-report tool that assesses the digital gaming attitude level. The lowest score that can be obtained from the scale is "18" and the highest score is "90". Change = ( Week 8 score - Baseline score).
Change from baseline in the 21-item Children's Self-Efficacy Scale score at 8 weeks. | Baseline and Week 8
  The Children's Self-Efficacy Scale is an approved self-report tool that assesses the level of self-efficacy. The lowest score that can be obtained from the scale is "21" and the highest score is "105". Change = ( Week 8 score - Baseline score).

CONTACTS AND LOCATIONS:
Overall Officials: Semra Zorlu, ass. prof., Study Director — Sivas Cumhuriyet Univercity
Locations (1):
- Amasya University, Amasya, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
sociodemographic data of the participants Results of the Digital Game Addiction Scale for Children Results of the Awareness Scale on Digital Gaming Addiction Digital Gaming Motivation Scale results Results of the Social Support Assessment Scale for Children and Adolescents Digital Gaming Attitude Scale results Results of the Self-Efficacy Scale for Children
Supporting Information: Study Protocol, ICF
Time Frame: 2 years
Access Criteria: The Council of Higher Education will be shared from the thesis center.
URL: https://tez.yok.gov.tr/UlusalTezMerkezi/giris.jsp

REFERENCES:
- [Derived] Memis A, Kocatas S. Effects of motivational interviews and hippotherapy on the digital game addiction levels of adolescents: Randomized controlled clinical trial. J Pediatr Nurs. 2025 Sep-Oct;84:133-141. doi: 10.1016/j.pedn.2025.05.024. Epub 2025 May 30. PMID 40449239